CLINICAL TRIAL: NCT06032156
Title: The Acute Effects of a High Versus Low Dose of a Ketone Monoester Supplement on Cerebral Blood Flow and Cognition
Brief Title: Ketone Dose and Cerebral Blood Flow Study
Acronym: kCBF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: kCBF
Record Dates: First submitted 2023-04-06; First posted 2023-09-11 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Cerebrovascular Function; Cognition
Keywords: Cerebral Blood Flow; Cognition; Beta-hydroxybutyrate (β-OHB)

STUDY DESIGN:
Intervention Model Description: A randomized double-blind placebo-controlled crossover design will be used to test 3 conditions. Participants will consume 60 mL of a supplement containing: 1) a low β-OHB dose (0.3g/kg) body weight of the ketone monoester; [R]-3-hydroxybutyl [R]-3-hydroxybutyrate); 2) a high β-OHB dose (0.6g/kg body weight); or 3) a taste-matched calorie-free inert placebo drink.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Single dose of a taste-matched calorie-free placebo
  Interventions: Other: Placebo
- High Dose β-OHB (Experimental): Single dose of a ketone monoester ([R]-3-hydroxybutyl [R]-3-hydroxybutyrate; 0.6 g β-OHB/kg body weight)
  Interventions: Dietary Supplement: High Dose β-OHB
- Low Dose β-OHB (Experimental): Single dose of a ketone monoester ([R]-3-hydroxybutyl [R]-3-hydroxybutyrate; 0.3 g β-OHB/kg body weight)
  Interventions: Dietary Supplement: Low Dose β-OHB

INTERVENTIONS:
Dietary Supplement: Low Dose β-OHB — Ingestion of a low dose [R]-3-hydroxybutyl [R]-3-hydroxybutyrate (0.3 g β-OHB/kg body weight) followed by 2-hours of rest. Submaximal exercise to be performed following 2-hour resting measures.
  Arms: Low Dose β-OHB
Dietary Supplement: High Dose β-OHB — Ingestion of a high dose [R]-3-hydroxybutyl [R]-3-hydroxybutyrate (0.6 g β-OHB/kg body weight) followed by 2-hours of rest. Submaximal exercise to be performed following 2-hour resting measures.
  Arms: High Dose β-OHB
Other: Placebo — Ingestion of a taste-matched calorie-free placebo drink followed by 2-hours of rest. Submaximal exercise to be performed following 2-hour resting measures.
  Arms: Placebo

SUMMARY:
Ketone bodies are produced by the liver during periods of food scarcity or severe carbohydrate restriction. Blood ketones are an alternative fuel source used by the brain, heart, and skeletal muscle during periods of fasting. Further, ketones bodies act as a signalling molecule that have pleiotropic effects that upregulate cellular stress-resistance pathways throughout the body.

Oral supplements containing exogenous ketones have recently become available and represent a novel tool for increasing plasma ketone bodies without the need for dietary restriction. Early evidence suggests that oral ketone supplements may enhance cerebral blood flow and improve cognition. However, the dose-dependent effects of a single ketone supplement on cerebral blood flow and cognition in young adults is currently unknown.

The purpose of this study is to characterize the effects of ingesting a high versus low dose of an oral ketone monoester on cerebral blood flow, circulating blood markers, and cognition in young adults.

As an exploratory aim, this study will investigate how oxygen uptake kinetics during submaximal exercise are impacted 2 hours after ingestion of a ketone supplement. Recent findings indicate that ketone supplementation may impair exercise performance due to the physiological stress (i.e., pH disturbances) imposed by an acute ketone dose. Delaying exercise onset by 2 hours after ingestion of a ketone supplement may enhance oxygen kinetics in a dose-dependent manner.

ELIGIBILITY:
Inclusion Criteria:

- Between the ages of 18 and 35

Exclusion Criteria:

* Presence of obesity (body mass index > 30 kg/m^2)
* Presence of known cardiovascular disease
* Presence of type 2 diabetes
* History of cardiovascular events requiring hospitalization (i.e., heart attack)
* History of concussion(s) with persistent symptoms
* Currently following a ketogenic diet and/or taking ketone body supplements

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Resting cerebral blood flow (CBF) | 2-hour
  Measured via duplex ultrasound of the extra-cranial arteries (internal carotid and vertebral arteries).

SECONDARY OUTCOMES:
Cognitive Function | 2-hour
  The MST (Mnemonic Similarity Task) will be used to assess hippocampal-dependent memory and pattern separation.
Plasma beta-hydroxybutyrate area under the curve | 2-hour
  Venous blood samples will be obtained via intravenous catheter
Brain-derived neurotrophic factor (BDNF) | 2-hour, then following completion of submaximal exercise bout
  Serum and plasma BDNF measured in venous blood samples will be obtained via intravenous catheter
Oxygen uptake (VO2) | 2-hour, then during submaximal exercise (performed after 2-hour rest period)
  Breath-by-breath analysis performed via metabolic cart
End-tidal CO2 | 2-hour, then during submaximal exercise (performed after 2-hour rest period)
  Breath-by-breath analysis performed via PowerLab Gas Analyzer (AD Instruments)
Mean arterial pressure (MAP) | 2-hour
  Automated blood pressure cuff measurement of brachial artery pressure in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy J Walsh, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon request
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Anyone who wishes to access the data.